CLINICAL TRIAL: NCT05285293
Title: Clinical Evaluation of Periodontal Regeneration Using Vitamin A Added to PRF in Comparison to PRF Alone in Treatment of Intra-bony Defects: Randomized Controlled Clinical Trial
Brief Title: Periodontal Regeneration Using Vitamin A and PRF Compared to PRF Alone Treating Intra-bony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdallah Hassan Mostafa, B.Sc., M.Sc. Abdallah Hassan Mostafa, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121221
Record Dates: First submitted 2022-03-03; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Intrabony Periodontal Defect
MeSH Terms: interventions — Prolactin-Releasing Hormone; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Control (Active Comparator): PRF in intra-bony defects
  Interventions: Biological: Platelet Rich Fibrin (PRF)
- Group 2 Experimental (Experimental): PRF and Retinol in intra-bony defects
  Interventions: Biological: Platelet Rich Fibrin (PRF) and Retinol

INTERVENTIONS:
Biological: Platelet Rich Fibrin (PRF) — Platelet rich fibrin (PRF) in treatment of intrabony defects using Modified Minimally invasive surgical technique (M-MIST)
  Arms: Group 1 Control
Biological: Platelet Rich Fibrin (PRF) and Retinol — Platelet rich fibrin (PRF) mixed with Retinol in treatment of intrabony defects using Modified Minimally invasive surgical technique (M-MIST)
  Arms: Group 2 Experimental

SUMMARY:
Will the addition of vitamin A (Retinol) to PRF add more periodontal regenerative value in the treatment of intra-bony defects compared to PRF alone, clinically?

DETAILED DESCRIPTION:
Vitamin A has been extensively studied for its role in bone health. Vitamin A can be consumed in two forms, i.e., preformed retinol and pro-vitamin A. Preformed retinol is often found in food originated from animals, such as dairy, liver and eggs. Provitamin A, such as alpha (α)-carotene, beta (β)-carotene orβ-cryptoxanthin, are commonly found in plant-based food, such as fruits and vegetables (Toti et al., 2018). At certain concentrations, it has been proven to enhance the pluripotency of periodontal cells for regeneration (Fawzy El-Sayed, Hein and Dörfer, 2019).

Yet, to the best of our knowledge no clinical trials have evaluated the effect of Vitamin A added to PRF in the regeneration of intra-bony defects. This study is to fill the gap of knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Stage III periodontitis patient (Papapanou et al., 2018) with 3 walled or 2 walled intra-bony defects.
* Non-smokers
* No pregnancy
* Medically free
* Presence of intra-bony defect of three or two walls (as predominant component) with a radiographic intra-bony component of ≥3 mm;
* Presence of ≥2 mm of keratinized gingiva at the tooth with the defect.
* Willingness to optimal compliance with the study procedures

Exclusion Criteria:

* Uncontrolled systemic or local infection in the tissue of interest,
* History or clinical evidence or positive tests for Human Immunodeficiency Virus (HIV), Hepatitis B virus (HBV), Hepatitis C virus (HCV).
* History of chronic autoimmune disease
* Participation in an intervention trial in the same quadrant in the previous two months.
* Type III tooth mobility, vertical root fracture in the selected tooth.
* Contraindications for periodontal surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic linear defect depth | 6 Month
  Measured as the depth of intra-osseous defect from the alveolar crest to the defect base (E et al., 2004)

SECONDARY OUTCOMES:
Clinical attachment level | 6 Month
  clinical attachment level measured in mm. using williams graduated probe(SP, 1967)
Probing pocket depth | 6 Month
  Measuring probing depth in mm using William's graduated Periodontal probe (SP, 1967)
Radiographic defect bone density | 6 MOnth
  Bone density will be measured using Digital Radiographs using ImageJ software (B et al., 2019)

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah H. Mostafa, M.Sc, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Inclusion, exclusion criteria, Methodology and Results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available once the study is over and for one year
Access Criteria: by emailing " Dr.abdallah.hassan@gmail.com"